CLINICAL TRIAL: NCT02103231
Title: Young Adult Cardiovascular Health sTudy
Acronym: YACHT
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: YACHT
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Preterm Birth; Hypertension
Keywords: Preterm birth; Hypertension; Exercise capacity; Cardiovascular risk
MeSH Terms: conditions — Premature Birth; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Full Term Birth: History of full term birth (>37 weeks gestation) including sub-group with diagnosis of hypertension
- Preterm Birth: History of preterm birth (<37 weeks gestation) including subgroup with diagnosis of hypertension

SUMMARY:
The purpose of this study is to understand more about why young people who were born prematurely may have increased risk of high blood pressure and lower cardiovascular exercise capacity.

DETAILED DESCRIPTION:
Young adults with a history of preterm birth are identified as having a unique risk profile for developing hypertension and having reduced exercise capacity. Globally, there are 15 million annual preterm births. In Europe, incidence is 6-15% of all births, with up to 6 million adults in the United Kingdom having a preterm birth history. Understanding the associations between early life exposures and this early cardiovascular risk is extremely important to be able to target primary prevention strategies.

As yet there are no clear explanations for the reduced exercise capacity and elevated risk of hypertension reported in preterm born young adults. Magnetic resonance imaging studies of young adult born premature demonstrated altered heart shape, with increased left ventricular mass, reduced cavity sizes and reduced stroke volumes. The changes in cardiac size identified from these studies is similar to those seen in other disease groups and has been equated to greater than 50% increased risk of cardiovascular clinical events in these groups. These structural changes may account for the reduced exercise capacity observed in preterm born young adults

This study aims to understand the physiological determinants of limited exercise capacity and associated cardiovascular risk profile of adult preterm born populations.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 to 40 years.
* History of preterm birth, diagnosis of hypertension or full term birth normotensive control
* Able (in the investigator's opinion) and willing to comply with all study requirements.
* Participant is freely able to access John Radcliffe Hospital for study visits

Exclusion Criteria:

* Aged <18 years >40 years
* Unwilling or unable to give informed consent for participation in the study.
* Pregnant or lactating during the course of the study.
* Planning to donate blood during the study duration.
* Any significant disease or disorder which, in the opinion of the investigator, might influence the participant's ability to participate in the study.
* Contraindication to Magnetic Resonance Imaging

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults aged between 18 and 40 years old, recruited from the local community and Oxford University Hospitals Hypertension clinic, participants will have a history of preterm (<37 weeks) or full term (>37 weeks) birth.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Capacity | Single measure, baseline study recruitment
  Peak oxygen uptake measured via cardiopulmonary exercise testing

SECONDARY OUTCOMES:
Cardiac Structure | Single measure, baseline recruitment
  Cardiac structure measured via cardiac magnetic resonance imaging
Cardiac Function | Single measure, baseline recruitment
  Cardiac function measured via cardiac magnetic resonance imaging
Liver Structure | Single measure, baseline recruitment
  Hepatic structure measured via magnetic resonance imaging
Brain structure | Second study visit within 6 months of recruitment
  Brain structure measured via magnetic resonance imaging
Vascular function | Single measure, baseline recruitment
  Vascular function measured via pulse wave velocity
Dynamic cardiac function | Single measure, baseline recruitment
  Dynamic cardiac function measured using echocardiogram during exercise

OTHER OUTCOMES:
Physical Activity Behaviour | Baseline recruitment
  Objective measure of physical activity using wrist worn accelerometer
Ambulatory Blood Pressure | Baseline Recruitment
  24 hour ambulatory blood pressure
Heart rate variability | Baseline measure
  24 hour heart rate variability
Microvascular measures | Single measure, baseline recruitment
  Capillary density measured using microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Paul Leeson, PhD, FRCP, Principal Investigator — University of Oxford Division of Cardiovascular Medicine; Adam J Lewandowski, DPhil, Study Director — University of Oxford Division of Cardiovascular Medicine
Locations (1):
- Adam Lewandowski, Oxford, England, United Kingdom

REFERENCES:
- [Derived] Mohamed A, Lamata P, Williamson W, Alsharqi M, Tan CMJ, Burchert H, Huckstep OJ, Suriano K, Francis JM, Pelado JL, Monteiro C, Neubauer S, Levy PT, Leeson P, Lewandowski AJ. Multimodality Imaging Demonstrates Reduced Right-Ventricular Function Independent of Pulmonary Physiology in Moderately Preterm-Born Adults. JACC Cardiovasc Imaging. 2020 Sep;13(9):2046-2048. doi: 10.1016/j.jcmg.2020.03.016. Epub 2020 May 13. No abstract available. PMID 32417327
- [Derived] Huckstep OJ, Williamson W, Telles F, Burchert H, Bertagnolli M, Herdman C, Arnold L, Smillie R, Mohamed A, Boardman H, McCormick K, Neubauer S, Leeson P, Lewandowski AJ. Physiological Stress Elicits Impaired Left Ventricular Function in Preterm-Born Adults. J Am Coll Cardiol. 2018 Mar 27;71(12):1347-1356. doi: 10.1016/j.jacc.2018.01.046. PMID 29566820